CLINICAL TRIAL: NCT04282902
Title: A Randomized, Open-label Study to Evaluate the Efficacy and Safety of Pirfenidone in Patients With Severe and Critical Novel Coronavirus Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of Pirfenidone With Novel Coronavirus Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huilan Zhang (Other)
Responsible Party: Sponsor-Investigator, Huilan Zhang, Associate Professor of department of respiratory and critical care medicine, tongji hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: huilanz_76
Record Dates: First submitted 2020-02-10; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Novel Coronavirus Pneumonia; Pneumonia; Pirfenidone
MeSH Terms: conditions — Pneumonia | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: This study planned to randomize approximately 147 adult subjects. They will be stratified according to whether the onset time is ≤14 days and randomly divided into groups of 1: 1, receiving standard treatment or pirfenidone orally 3 times a day, 2 tablets each time. The course is 4 weeks or more. Subjects and all research center staff were not blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): This study was designed to randomize approximately 147 adult subjects.The patients were stratified according to whether the onset time was less than 14 days, and randomly divided into groups at a ratio of 1:1. The group received pirfenidone orally three times a day, with two tablets each time, for a course of 4 weeks or longer.
  Interventions: Drug: pirfenidone
- Standard treatment group (No Intervention): This study planned to randomize approximately 147 adult subjects. They will be stratified according to whether the onset time is ≤ 14 days and randomly divided into groups of 1: 1. This group only receives standard treatment

INTERVENTIONS:
Drug: pirfenidone — Pirfenidone is administered orally 3 times a day, 2 tablets each time, for a period of 4 weeks or longer
  Arms: Pirfenidone group

SUMMARY:
The acute lung injury caused by SARS and 2003 were both related to the inflammatory cytokine storm in patients. The biochemical test showed abnormal increase in related indicators such as interleukin-8, and CT images showed a medical "white" lung". According to the experience of SARS treatment in 2003, the use of hormones will indeed help the patients to alleviate their illness, but patients who survived SARS either had too much hormone at that time and took too long. Although the lungs could recover, but the femoral head was necrotic Either the amount of hormones was very conservative at the time, which kept the lungs in the storm of inflammatory factors, leading to the emergence of irreversible pulmonary fibrosis. So is there a medicine that can anti-inflammatory, reduce the load of hormone use, and have the effect of treating and preventing pulmonary fibrosis complicated by severe viral lung? At present, pirfenidone has achieved encouraging results in the treatment of idiopathic Pulmonary Fibrosis (CTD-ILD) diseases. It is particularly encouraging that the values announced at the 2019 ATS Annual Conference suggest that pirfenidone has more anti-inflammatory and anti-oxidant effects than its own outstanding anti-fibrotic ability. The data shows early use, Its strong anti-SOD activity can effectively inhibit IL-1beta and IL-4, and can open the prevention mode of pulmonary interstitial fibrosis. Based on the above, this project intends to make the following scientific assumptions: based on the homology of the pathogens of the new coronavirus-infected pneumonia and the coronavirus infection of pneumonia in 2003, the similarities in the occurrence and development of the disease, that is, the pulmonary inflammatory storm occurs first, and thereafter The progress of fibrosis and the progressive decline of lung function and mortality are higher than those of ordinary pneumonia. We hope that by adding pirfenidone as a treatment program in addition to standard treatment, it will be a new and severe type of coronavirus infection. Patient clinical treatment provides an effective and practical method.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open, blank-controlled, multi-stage clinical study. As there are no effective treatments, the project team will evaluate possible treatments (including but not limited to Pirfenidone) based on actual conditions. Ketone, Pirfenidone, lopinavir / ritonavir, remdesivir, single / polyclonal antibodies against coronavirus), explore the most effective treatment options.

The first phase will assess the efficacy and safety of approximately 147 (primarily estimated) hospitalized adult patients diagnosed with Wuhan new coronavirus infection in the pirfenidone-treated group compared to standard treatment.

Patients with influenza within 14 days of onset of symptoms were screened and randomly assigned as soon as possible after screening (within 4 day). Patients will be allocated in a 1: 1 ratio and divided into the pirfenidone treatment group or the standard treatment group only. Patients who do not meet the inclusion and exclusion criteria are only allowed to be re-screened once, provided that the time from onset of symptoms to randomization remains within 14days.

This study planned to randomize approximately 147 adult subjects. They will be stratified according to whether the onset time is ≤ 14 days and randomly divided into groups of 1: 1, receiving standard treatment or pirfenidone orally 3 times a day, 2 tablets each time. The course is 4 weeks or more. Subjects and all research center staff were not blinded.

Study selection criteria: (1) Age ≥ 18 years. (2) Clinically diagnosed patients with new type of coronavirus pneumonia include: on the basis of meeting the criteria for suspected cases, one of the following pathogenic evidence: ① real-time fluorescent RT-PCR of respiratory specimens or blood specimens for detection of new coronavirus nucleic acid; Respiratory or blood specimens are genetically sequenced and highly homologous to known new coronaviruses. (3) The time interval between the suspected neocoronary pneumonia pneumonia case and the random enrollment is determined within 4 days to 7 days according to the history symptoms and chest CT imaging. Cough, diarrhea, or other related symptoms can be used. The imaging changes are mainly based on chest CT.

Study exclusion criteria: (1) AST and ALT> 1.5 x ULN at visit 1; (2) bilirubin> 1.5 x ULN at visit 1; (3) Cockcroft-Gault formula at visit 1 Calculated creatinine clearance rate <30 mL / min; (4) patients with potential chronic liver disease (Child Pugh A, B or C liver injury; (5) previous treatment with nidanib or pirfenidone; Screening visit (Visit 1) 1 month or 6 half-life (whichever is greater) received other research drug treatment; (7) Based on ATS / ERS / JRS / ALAT 2011 guidelines (P11-07084) IPF diagnosis; (8) Obvious pulmonary hypertension (PAH) defined by any of the following standards: ① Clinical / echocardiographic evidence of previously obvious right heart failure; ② Medical history including right heart catheter showing a heart index ≤ 2l / min / m2; ③ required Parenteral administration of epoprostenol / treprostinil for the treatment of PAH; (9) other clinically significant pulmonary abnormalities considered by the investigator; (10) major extrapulmonary physiological limitations (such as chest wall deformities, large amounts Pleural effusion); (11) cardiovascular disease, any of the following diseases: ① severe hypertension within 6 months of visit 1, treatment Uncontrollable (≥160 / 100 mmHg); ② myocardial infarction within 6 months of visit 1; ③ unstable angina within 6 months of visit 1; (12) history of severe central nervous system (CNS) events; (13) Known allergies to the test drug; (14) Other diseases that may interfere with the testing process or judged by the investigator may interfere with the trial participation or may put the patient at risk when participating in the trial; (15) pregnancy, Women who are breastfeeding or planning a pregnancy; (16) Patients are unable to understand or follow the test procedures, including completing the questionnaires themselves without help.

Study design primary and secondary endpoints Main endpoints: (1) Absolute changes in baseline lesion area, finger pulse oxygen, and blood gas from baseline at 4 weeks of chest CT images; (2) Total score of King's Interstitial Lung Disease Short Questionnaire (K-BILD) at Week 4 Absolute change from baseline.

Secondary end point: Time to death within 4 weeks due to respiratory causes; time to disease progression or death within 4 weeks; recovery of blood routine lymphocytes at week 4; and blood inflammation indicators at week 4 ( IL-8, etc.); at week 4, absolute changes in viral nucleic acid from baseline; at week 4, pulmonary fibrosis survival symptoms dyspnea scores absolute changes from baseline; at week 4, pulmonary fibrosis survival Symptoms of cough scores are absolute changes from baseline.

ELIGIBILITY:
Inclusion Criteria:

(1) Age ≥ 18 years. (2) Clinically diagnosed patients with new type of coronavirus pneumonia include: on the basis of meeting the criteria for suspected cases, one of the following pathogenic evidence: ① real-time fluorescent RT-PCR of respiratory specimens or blood specimens for detection of new coronavirus nucleic acid; Respiratory or blood specimens are genetically sequenced and highly homologous to known new coronaviruses. (3) The time interval between the suspected neocoronary pneumonia pneumonia case and the random enrollment is determined within 4 days to 7 days according to the history symptoms and chest CT imaging. Cough, diarrhea, or other related symptoms can be used. The imaging changes are mainly based on chest CT.

Exclusion Criteria:

(1) AST and ALT> 1.5 x ULN at visit 1; (2) bilirubin> 1.5 x ULN at visit 1; (3) creatinine clearance rate calculated by Cockcroft-Gault formula at visit 1 <30 mL / min; (4) patients with potential chronic liver disease (Child Pugh A, B or C liver injury; (5) previous treatment with nidanib or pirfenidone; (6) screening visits (interviews 1) Received other research drug treatment within 1 month or 6 half-lives (whichever is greater); (7) IPF diagnosis based on ATS / ERS / JRS / ALAT 2011 guidelines (P11-07084); (8 ) Significant pulmonary hypertension (PAH) defined by any of the following standards: ① Clinical / echocardiographic evidence of previously significant right heart failure; ② Medical history including right heart catheter showing a cardiac index ≤ 2l / min / m2; ③ Prostaglandol / qu Parenteral administration of prostacyclin in the treatment of PAH; (9) other clinically significant lung abnormalities considered by the investigator; (10) major extrapulmonary physiological limitations (such as chest wall deformity, large amount of pleural effusion); (11) Cardiovascular diseases, any of the following diseases: ① Severe hypertension within 6 months of Visit 1, uncontrollable after treatment (≥160 / 100 mmHg); ② myocardial infarction within 6 months of visit 1; ③ unstable angina within 6 months of visit 1; (12) history of severe central nervous system (CNS) events; (13) known trials Drug allergies; (14) Other diseases that may interfere with the testing process or as judged by the investigator may interfere with the trial participation or may put the patient at risk when participating in the trial; (15) Women who are pregnant, breastfeeding, or planning pregnancy in this trial (16) Patients are unable to understand or follow the trial procedures, including completing the questionnaires themselves without assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
chest CT | 4 weeks
  Lesion area of chest CT image at 4 weeks
Finger pulse oxygen | 4 weeks
  Absolute change in pulse oxygen from baseline
blood gas | 4 weeks
  Absolute change in blood gas from baseline
K-BILD | 4 weeks
  Absolute change in total score of King's brief questionnaire for interstitial Absolute change in total score of King's brief questionnaire for interstitial pulmonary disease (k-bild) from baseline at week 4

SECONDARY OUTCOMES:
death | 4 weeks
  Time to death within 4 weeks due to respiratory problems
Time to disease progression or death within 4 weeks | 4 weeks
  Time to disease progression or death within 4 weeks
blood | 4 weeks
  lymphocyte count
viral nucleic acid | 4 weeks
  Absolute change in viral nucleic acid from baseline
dyspnea score | 4 weeks
  Pulmonary fibrosis survival symptoms absolute changes in dyspnea score from baseline
blood | 4 weeks
  changes in blood inflammatory indexes
cough scores | 4 weeks
  Absolute change in cough scores for pulmonary fibrosis survival symptoms from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital affiliated to huazhong university of science and technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dewage SNV, Organ L, Koumoundouros E, Derseh HB, Perera KUE, Samuel CS, Stent AW, Snibson KJ. The efficacy of pirfenidone in a sheep model of pulmonary fibrosis. Exp Lung Res. 2019 Nov-Dec;45(9-10):310-322. doi: 10.1080/01902148.2019.1695019. Epub 2019 Nov 25. PMID 31762329
- [Result] Lehmann M, Buhl L, Alsafadi HN, Klee S, Hermann S, Mutze K, Ota C, Lindner M, Behr J, Hilgendorff A, Wagner DE, Konigshoff M. Differential effects of Nintedanib and Pirfenidone on lung alveolar epithelial cell function in ex vivo murine and human lung tissue cultures of pulmonary fibrosis. Respir Res. 2018 Sep 15;19(1):175. doi: 10.1186/s12931-018-0876-y. PMID 30219058
- [Result] Ikeda S, Sekine A, Baba T, Katano T, Tabata E, Shintani R, Sadoyama S, Yamakawa H, Oda T, Okuda R, Kitamura H, Iwasawa T, Takemura T, Ogura T. Negative impact of anorexia and weight loss during prior pirfenidone administration on subsequent nintedanib treatment in patients with idiopathic pulmonary fibrosis. BMC Pulm Med. 2019 Apr 11;19(1):78. doi: 10.1186/s12890-019-0841-7. PMID 30975118
- [Result] Epstein Shochet G, Wollin L, Shitrit D. Fibroblast-matrix interplay: Nintedanib and pirfenidone modulate the effect of IPF fibroblast-conditioned matrix on normal fibroblast phenotype. Respirology. 2018 Aug;23(8):756-763. doi: 10.1111/resp.13287. Epub 2018 Mar 12. PMID 29532550